CLINICAL TRIAL: NCT03327519
Title: Solving Insomnia Electronically: Sleep Treatment for Asthma
Acronym: SIESTA
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: issue reaching target enrollment
Sponsor: University of Pittsburgh (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Faith Luyster, Associate Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRO17040267; R01HL131587-01A1 (NIH)
Record Dates: First submitted 2017-10-26; First posted 2017-10-31 (Actual); Last update posted 2023-07-21 (Actual); Status verified 2023-07

CONDITIONS: Asthma; Insomnia
Keywords: Asthma; Insomnia
MeSH Terms: conditions — Asthma; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: experimental, longitudinal, randomized controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- SHUTi (Experimental): Self-guided, automated, interactive, and tailored web-based program
  Interventions: Behavioral: SHUTi
- Emmi (Experimental): A program that is an animated online video that walks patients through important information about a health topic, condition or procedure.
  Interventions: Behavioral: Emmi

INTERVENTIONS:
Behavioral: SHUTi — Sleep Healthy Using the Internet (SHUTi) is a self-guided, automated, interactive, and tailored web-based program modeled on the primary tenets of CBT-I: sleep restriction, stimulus control, cognitive restructuring, sleep hygiene, and relapse prevention.
  Arms: SHUTi
Behavioral: Emmi — The Emmi® program for insomnia contains educational information on physiological controls of sleep, sleep hygiene practices, healthy sleep behaviors (e.g., reduce time in bed, get up at the same time every day, go to bed only if sleepy, and do not stay in bed unless asleep), and sleep medications; assesses self-efficacy, and; allows patients to set individual goals.
  Arms: Emmi

SUMMARY:
Insomnia is commonly reported by adults with asthma. Insomnia can worsen asthma patients' quality of life and increase the risk for asthma attacks.This clinical trial will compare sleep and asthma control in adults with asthma and insomnia who receive either an internet-based intervention for insomnia or an educational video about insomnia.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 years
2. Telephone, email address, reliable Internet access
3. Have a current primary care physician or a physician who is managing patient's asthma
4. Diagnosis of asthma supported by at least one of the following:

   1. Patient self-report of physician diagnosis of asthma
   2. Asthma diagnosis in the electronic medical record
5. Self-report of current use of medications for asthma
6. FEV1 of ≥ 45% of the predicted normal value for the patient, after withholding bronchodilators at or personal best peak expiratory flow of > 100 L/min
7. Not well-controlled asthma: Score 12-19 on Asthma Control Test for those on an inhaled corticosteroid; Score 16-19 on Asthma Control Test for those not on an inhaled corticosteroid.
8. Impaired asthma-specific quality of life: Score ≤ 5 on Asthma Quality of Life Questionnaire
9. If subjects are on a controller medication (i.e., inhaled corticosteroid, inhaled corticosteroid and long acting beta-agonists, Singulair, etc.), they must be on stable doses and schedules (i.e., unchanged) of therapy for 2 months prior to enrollment.
10. Meets criteria for DSM-5 Insomnia Disorder
11. At least moderate insomnia severity: Score > 7 on Insomnia Severity Index
12. Stable self-reported medical, psychiatric conditions

Exclusion Criteria:

1. Non-English speaking, illiterate, or sensory deficits
2. Plans to move or leave present source of care during the following 8 months
3. Receiving antibiotics for upper respiratory infection or pulmonary condition in previous 2 weeks
4. Heavy smoking: Age < 30 years and smoking history > 10 pack years OR age ≥ 30 and smoking history > 15 pack years OR smoking within previous 12 months
5. Substance abuse disorder within previous 3 months
6. Self-reported cystic fibrosis, COPD or interstitial lung disease
7. Self-report of > 3 asthma attacks/exacerbations requiring systemic corticosteroids, emergency room visit, or hospitalization within the previous year
8. Oral corticosteroid dosage of > 10 mg/daily
9. Poorly controlled gastroesophageal reflux disease (GERD)
10. Untreated severe obstructive sleep apnea based on apnea-hypopnea index of ≥ 55
11. Self-reported untreated restless legs syndrome
12. History of bipolar disorder or psychosis
13. Current major depression or active suicidal ideation.
14. Asthma attacks/exacerbations requiring systemic corticosteroids, emergency room visit, or hospitalization within the previous 4 weeks
15. Self-report of current pregnancy or trying to become pregnant. Participants who become pregnant during course of the study will be withdrawn from the study.
16. Shift work that includes working the night shift (between the hours of 12:00 a.m. - 6:00 a.m.)
17. Enrolled in prior R03 study (HL135213)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2018-05-29 (Actual); Primary Completion 2022-08-15 (Actual); Study Completion 2022-08-15 (Actual)

PRIMARY OUTCOMES:
The Insomnia Severity Index (ISI) | Change from Baseline to 3 & 6 months from start of intervention
  The Insomnia Severity Index is a 7-item self-report questionnaire assessing nature, severity and impact of insomnia symptoms. The total score ranges from 0 to 28, with higher scores indicating worse insomnia severity.

SECONDARY OUTCOMES:
Asthma Quality of Life Questionnaire (AQLQ) | Change from Baseline to 3 & 6 months from start of intervention
  The Asthma Quality of Life Questionnaire is a 32-item measure assessing asthma-specific health-related quality of life in 4 domains: activity limitations (ability to carry out daily activities), symptoms (frequency and nature of asthma symptoms such as coughing and chest tightness), emotional distress (intensity of the discomfort, fear, or distress associated with asthma), and environmental stimuli (capacity to manage environmental triggers of asthma such as smoke, dust, and pollution). An overall total score is computed by averaging the scores from the four domains. The total score ranges from 1 to 7, with higher scores indicating better quality of life.
Asthma Control Test (ACT) | Change from Baseline to 3 & 6 months from start of intervention
  The Asthma Control Test is a 5-item questionnaire that measures asthma control by assessing interference with activity, shortness of breath, nocturnal symptoms, rescue medication use, and self-rating of asthma control. The total score ranges from 5 to 25, with higher scores indicating greater asthma control.

CONTACTS AND LOCATIONS:
Overall Officials: Faith Luyster, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh Asthma Insititute @ UPMC, Pittsburgh, Pennsylvania, United States